CLINICAL TRIAL: NCT04492956
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Exploratory Study to Evaluate the Efficacy and Safety of Ecopipam Tablets in Adults With Childhood Onset Fluency Disorder (Stuttering)
Brief Title: Effects of Ecopipam or Placebo in Adults With Stuttering (Speak Freely)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: University of California, Riverside (Other); Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBS-101-COFD-201
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Childhood-Onset Fluency Disorder (Stuttering)
Keywords: Stuttering; Communication Disorders
MeSH Terms: conditions — Childhood-Onset Fluency Disorder; Stuttering; Communication Disorders | interventions — ecopipam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ecopipam HCl ~2mg/kg/day (Experimental): Ecopipam HCl tablets of 12.5, 50, and 75 mg for daily, oral administration for 12 weeks
  Interventions: Drug: Ecopipam
- Matching Placebo (Placebo Comparator): Matching placebo tablets for daily, oral administration for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecopipam — Oral tablet
  Arms: Ecopipam HCl ~2mg/kg/day
Drug: Placebo — Oral tablet
  Arms: Matching Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, Phase 2 exploratory study in adult subjects with childhood onset fluency disorder.

DETAILED DESCRIPTION:
At the Baseline visit, eligible subjects will be randomized 1:1 to receive either a target steady-state dose of ecopipam HCl ~2 mg/kg/day or matching placebo for a 12-week Treatment Period consisting of a 4-week Titration Phase followed by an 8-week Maintenance Phase.

Subjects will return to the clinic at 4, 8, and 12 weeks after Randomization and Follow-up visits 7 and 14 days after completing the Treatment Period or Early Discontinuation. Efficacy assessments will be conducted at Weeks 4, 8, and 12 and safety assessments will be conducted at all visits. Subjects will have adverse events and other safety parameters assessed by phone or video conference at Weeks 2, 6 and 10 and 30 days after the last study drug administration. Signs or symptoms of withdrawal, abuse, and dependence will be monitored throughout the study.

At the end of the Treatment Period or Early Discontinuation, subjects will taper study drug by 25 mg/day until off study drug, for up to 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in English and provide informed consent
* 18 years or older of age at screening
* Weighs >= 45 kg (~99 lbs)
* Satisfies DSM-5 criteria for childhood onset fluency disorder
* History of stuttering for >=2 years with onset consistent to developmental in nature
* Must meet an allowed severity of stuttering at screening and baseline, scored by a central rater
* Completed an adequate course of speech therapy
* Has a qualifying IOS or Android smartphone
* Must discontinue all medications used to treat stuttering for at least 14 days prior to screening
* Sexually active females of child bearing potential must be using effective contraception during and 30 days after participation
* Sexually active males must use a double barrier method of contraception during and 30 days after participation

Exclusion Criteria:

* Stuttering is related to a known neurological cause
* Initiation of new behavioral therapies for stuttering within 10 weeks prior to baseline
* Unstable medical illness or clinically significant abnormalities on screening tests/exams
* At a significant risk of committing suicide
* Are pregnant or lactating
* Positive urine drug screen
* Lifetime history of major depressive episode
* History of seizures
* Have been previously treated with ecopipam
* Unstable use of medications prior to screening
* Use of prohibited medications or need for medications which would have unfavorable interactions with ecopipam
* Not suitable for study in the opinion of the Principle Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Stuttering Severity Instrument, 4th edition (SSI-4) baseline to Week 12 | 12 weeks
  Measures stuttering severity in children and adults

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) baseline to Week 12 | 12 weeks
  Rates the severity of the subject's illness at the time of assessment, relative to the the clinician's past experience with patients who have the same diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Atul R Mahableshwarkar, MD, DFAPA, Study Director — Emalex Biosciences Inc.
Locations (9):
- United States (9):
  - UC Riverside, Riverside, California
  - CI Trials, Santa Ana, California
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - Institute For Advanced Medical Research, Atlanta, Georgia
  - Social Psychiatry Research Institute, Prairie Village, Kansas
  - Michigan State University, East Lansing, Michigan
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Clinical Neuroscience Solutions Inc, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No